CLINICAL TRIAL: NCT04988724
Title: Impact of Physical Exercise at a Hospital Tested in a Pilot Trial
Brief Title: Impact of Physical Exercise at a Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Stig Molsted, Associate Professor, Nordsjaellands Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-21021866
Record Dates: First submitted 2021-06-29; First posted 2021-08-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pain; Quality of Life; Health Behavior
MeSH Terms: conditions — Pain; Health Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pilot study without control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Intervention group that receive 30 min exercise training twice weekly in 20 weeks
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Exercise training with aerobic and strength training, 30 min per session

SUMMARY:
Aims and Hypotheses Aims

* to investigate associations between an intelligent exercise training intervention and clinical health parameters, well-being, sick leave and productivity at Nordsjællands Hospital (NOH)
* to generate data and experiences to a larger cluster randomized trial with more included departments at NOH
* to analyze how the intervention could be successfully implemented in the organization to ensure long-term effects

Outcomes

* Aerobic capacity (Åstrand's ergometer test)
* Blood pressure and heart rate
* Physical activity (steps measured by tracker)
* Self-reported health (questionnaire EQ-5D)
* Self-reported physical activity (questionnaire IPAQ)
* Well-being (questions from the Danish Health and Morbidity Survey)
* Musculoskeletal pain and use of anti-pain medications (Numeric Rating Scale)
* Monetized value of productivity loss
* Productivity using an employer´s perspective (scale 1-10)
* Sick leave (days in short term (≤14 days) and long term (>14 days), data will be delivered by The Department of HR)
* Muscle strength in knee extension (dynamometer)

Intervention The concept of intelligent training at the worksite is an individualized exercise training where the exercises are: 1) balanced to the physiological capacity of the employees relative to their occupational exposure, 2) tailored to the individual capacities and disorders to improve employees' health, 3) motivating by offering evidence based and enjoyable programs implemented with care, and 4) cost-effective for the company.

The intervention period is 20 weeks of intelligent exercise training. Every week, several exercise sessions will be offered to the participants in the intervention group during the working hours. The exercise sessions will be of 30 min durations twice a week and include aerobic exercise with high intensity (≥16 on the Borg scale, rate of perceived exhaustion), resistance training and/or functional training. In addition, there will be a number of intelligent exercise sessions of 30 min durations before and after the most common working hours with a primary focus on aerobic exercise. The exercise sessions will be supervised by exercise experts (education in sport or physiotherapy).

The intelligent exercise interventions will be adjusted to the individual participant's physical capacity and limitations; thus, as one participant may perform aerobic exercise, another person may perform resistance training.

DETAILED DESCRIPTION:
In this pilot study, we will investigate the potential of physical training at departments at NOH. A large university hospital covering a population of 1,7 mio citizens in the Northern Region of Zealand, and one of eight new Danish "super-hospitals". We will invite all health care workers from the participating departments at the hospital to be enrolled in the study and apply the "intelligent exercise" intervention where each participant will receive a tailored intervention (exercise plan) based on an individual assessment including the mapping of the participant's needs and motivation (2).

References can be found at the end of the document.

Participants The 15 departments will be invited and it is anticipated that 700 employed will volunteer to the study.

All employees (nurses, doctors, secretaries and other staff) in the departments will be invited to the study. The recruitment will follow a strategy with local information at the departments regarding the study intervention and tests.

Intervention The concept of intelligent training at the worksite is an individualized exercise training where the exercises are: 1) balanced to the physiological capacity of the employees relative to their occupational exposure, 2) tailored to the individual capacities and disorders to improve employees' health, 3) motivating by offering evidence based and enjoyable programs implemented with care, and 4) cost-effective for the company.

The intervention period is three months of intelligent exercise training. Every week, several exercise sessions will be offered to the participants in the intervention group during the working hours. The exercise sessions will be of 30 min durations twice a week and include aerobic exercise with high intensity (≥16 on the Borg scale, rate of perceived exhaustion), resistance training and/or functional training (12). In addition, there will be a number of intelligent exercise sessions of 30 min durations before and after the most common working hours with a primary focus on aerobic exercise. The exercise sessions will be supervised by exercise experts (education in sport or physiotherapy).

The intelligent exercise interventions will be adjusted to the individual participant's physical capacity and limitations; thus, as one participant may perform aerobic exercise, another person may perform resistance training (12).

A goal will be that as many as possible will participate in minimum 60 min intelligent exercise training per week.

Prior to the intervention the participants will also be offered motivational support by a special educated staff to increase the level of leisure time physical activity and the level of general physical activity at work.

There will be offered intelligent exercise interventions to those on evening duties.

During the intervention periods, the participants will be supported by trained exercise ambassadors.

Sample size calculation The study will be performed without a sample size calculation, as it is a pilot trial to generate data before the intervention is tested in a larger cluster randomized trial with sufficient power to assess the validity of the results.

Statistical analyses The analyses of the changes of the numeric outcome variables during the study will be assessed using Student's t test if data are normally distributed or Wilcoxon Signed Ranks Test if data are not normally distributed. Changes of categorical variables will be analysed using a Chi2 test.

The associations between groups of staff (nurses, medical doctors and other) and changes of outcome variables (physical activity, productivity, sick leave, physical capacity) will be tested in multiple linear regression models with confounder adjustments.

Results are considered significant (2-tailed) when p<0.05. The statistical analyses will be performed in collaboration with a statistician from Section of Biostatistics, Department of Public Health, University of Copenhagen.

Subjects Every employee (e.g. nurses, doctors, secretaries, lab technician) from the departments at NOH will be invited to the study, but only those who agree in writing will be included.

Short-term and long-term risks, side effects and disadvantages Participants who have not previously been physically active may experience transient side effects such as sore muscles, shortness of breath, etc. There are no immediate risks associated with the intervention, as it is adapted to the physical ability of the individual subject. The therapeutic benefit for participants and future employees justifies an intervention like this.

Biological material None

Processing of personal data in the project The study will be approved by the Danish Data Protection Agency. The collected data will be stored in RedCap according to rules of the data protection agency in the Capital Region. All project data collected, will be handled in accordance with the rules of the Capital Region, in relation to current legislation. No data are sent abroad.

Funding The initiative to plan and execute the study is done by senior researcher associate professor Stig Mølsted and other researchers employed at NOH. The study is supported by NOH with a grant of 50,000 DKK to the initial analysis. In addition, NOH supports the study with other payments including the costs related to the participants' exercise training during the working hours. To ensure the realizability of this study, several funding application initiatives are in the pipeline for 2021-3 and forth, including Danish national and private funds.

Grants will be deposited into a hospital account. Members of the study group will have no financial affiliation with donors.

Remuneration No remuneration is paid to the project participants

Recruitment of subjects and informed consent Potential study participants in the included departments will receive written information about the project explaining the intervention. Oral information will be provided at joint meetings at the hospital to which test subjects are invited. Interested participants will also receive a written consent form. Prior to obtaining the informed consent, it will be ensured that the participants will have time and opportunity to read the information, ask questions and consider whether to participate. If the participant wishes to be included in the study, the consent declaration is dated and signed by the study participant and by the health care professional who provided the information.

Presentation of the results The results should have special interest to hospitals in Denmark and worldwide. The results of the study will also be of interest in other public and private companies.

The study results will be presented at national and international meetings and congresses, in international peer reviewed journals and in public media. Both positive, negative and inconclusive results will be published. The study will be registered at www.clinicaltrials.gov.

Ethics In this scientific experiment, all participants receive a training program tailored to the individual. Each individual participant is being physically pressured to an extent that one must not assume will be of any long-term burden to the participant. If any test results call for further investigations of a participant, the participant will be encouraged to consult the person's general practitioner.

Adverse effects related to the exercise interventions will be registered and evaluated in the study. The therapeutic benefit for participants and future employees justifies an intervention like this, as this intervention is expected to raise public health in general.

Adverse effects related to the exercise interventions will be registered and evaluated in the study.

References

1. Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports 2015 Dec;25 Suppl 3:1-72.
2. Justesen JB, Sogaard K, Dalager T, Christensen JR, Sjogaard G. The Effect of Intelligent Physical Exercise Training on Sickness Presenteeism and Absenteeism Among Office Workers. J Occup Environ Med 2017 Oct;59(10):942-948.
3. Jakobsen MD, Sundstrup E, Brandt M, Andersen LL. Psychosocial benefits of workplace physical exercise: cluster randomized controlled trial. BMC Public Health 2017 Oct 10;17(1):798-017-4728-3.
4. Korshoj M, Birk Jorgensen M, Lidegaard M, Mortensen OS, Krustrup P, Holtermann A, et al. Decrease in musculoskeletal pain after 4 and 12 months of an aerobic exercise intervention: a worksite RCT among cleaners. Scand J Public Health 2018 Dec;46(8):846-853.
5. Blangsted AK, Sogaard K, Hansen EA, Hannerz H, Sjogaard G. One-year randomized controlled trial with different physical-activity programs to reduce musculoskeletal symptoms in the neck and shoulders among office workers. Scand J Work Environ Health 2008 Feb;34(1):55-65.
6. Jakobsen MD, Sundstrup E, Brandt M, Jay K, Aagaard P, Andersen LL. Effect of workplace- versus home-based physical exercise on musculoskeletal pain among health care workers: a cluster randomized controlled trial. Scand J Work Environ Health 2015 Mar;41(2):153-163.
7. van den Berg S, Burdorf A, Robroek SJW. Associations between common diseases and work ability and sick leave among health care workers. Int Arch Occup Environ Health 2017 Oct;90(7):685-693.
8. European Foundation for the Improvement of Living and Working Conditions. http://www.eurofound.europa.eu/. Absence from work. © European Foundation for the Improvement of Living and Working Conditions, 2010.
9. Korshoj M, Lidegaard M, Skotte JH, Krustrup P, Krause N, Sogaard K, et al. Does aerobic exercise improve or impair cardiorespiratory fitness and health among cleaners? A cluster randomized controlled trial. Scand J Work Environ Health 2015 Mar;41(2):140-152.
10. Lidegaard M, Sogaard K, Krustrup P, Holtermann A, Korshoj M. Effects of 12 months aerobic exercise intervention on work ability, need for recovery, productivity and rating of exertion among cleaners: a worksite RCT. Int Arch Occup Environ Health 2018 Feb;91(2):225-235.
11. Andersen LL, Kjaer M, Sogaard K, Hansen L, Kryger AI, Sjogaard G. Effect of two contrasting types of physical exercise on chronic neck muscle pain. Arthritis Rheum 2008 Jan 15;59(1):84-91.
12. Sjogaard G, Justesen JB, Murray M, Dalager T, Sogaard K. A conceptual model for worksite intelligent physical exercise training--IPET--intervention for decreasing life style health risk indicators among employees: a randomized controlled trial. BMC Public Health 2014 Jun 26;14:652-2458-14-652.
13. Danish Health and Medicines Authority. [Specialeplanlægning]. 2015 April;978-87-7104-601-4(1.1).
14. Danmarks Radio. [Danmarkskort: Her er der størst lægemangel]. 2018; Available at: https://www.dr.dk/nyheder/indland/danmarkskort-her-er-der-stoerst-laegemangel. Accessed 08.29., 2019.
15. Kristensen MT. [Sundhedsreform kan forværre manglen på prkatiserende læger, hvor den er størst]. 2019(10).
16. Danmarks Radio. [Lægemangel i uskantsområderne er tredoblet under Lars Løkke]. 2019; Available at: https://www.dr.dk/nyheder/politik/laegemangel-i-udkantsomraaderne-er-tredoblet-under-lars-loekke. Accessed 08.29., 2019.
17. Pronk NP, Martinson B, Kessler RC, Beck AL, Simon GE, Wang P. The association between work performance and physical activity, cardiorespiratory fitness, and obesity. J Occup Environ Med 2004 Jan;46(1):19-25.
18. Pereira M, Comans T, Sjogaard G, Straker L, Melloh M, O'Leary S, et al. The impact of workplace ergonomics and neck-specific exercise versus ergonomics and health promotion interventions on office worker productivity: A cluster-randomized trial. Scand J Work Environ Health 2019 Jan 1;45(1):42-52.
19. Jensen TM, Eriksen SBM, Larsen JS, Aadahl M, Rasmussen SS, Olesen LB, et al. Exercise training is associated with reduced pains from the musculoskeletal system in patients with type 2 diabetes. Diabetes Res Clin Pract 2019 154:124-129.

ELIGIBILITY:
Inclusion Criteria:

- Employed nurses, doctors, secretaries and other staff on Nordsjællands Hospital, Denmark

Exclusion Criteria:

- If exercise training is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-04-16 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of work productivity | Tested before and after 20 weeks intervention
  Self-rated in questionaire (1-10 scale)

SECONDARY OUTCOMES:
Changes of personal well-being | Tested before and after 20 weeks intervention
  Self-rated in questionaire (likert scale)
Changes of quality of life | Tested before and after 20 weeks intervention
  Self-rated quality of life in the questionaire EQ-5D (scale -0.624 to 1)
Changes in self-rated physical activity | Tested before and after 20 weeks intervention
  Self-rated in the questionaire IPAQ (total METs scores, continous data)
Changes of muscoloskeletal pain | Tested before and after 20 weeks intervention
  Self-rated in questionaire (NRS 0-10)
Changes of blood pressure | Tested before and after 20 weeks intervention
  Resting test of diastolic and systolic pressure (mmHg)
Changes of aerobic capacity | Tested before and after 20 weeks intervention
  Aastrands test (oxygen uptace pr min pr kg body weight)
Changes of hip/waist ratio | Tested before and after 20 weeks intervention
  The circumferences of the hip and waist areas (cm)
Changes of sick-leave | Tested before and after 20 weeks intervention
  Register data for sick-leave (number of days)
Changes of physical activity | Tested before and after 20 weeks intervention
  Tracked by telephones (health app, number of steps)
Changes of muscle strength | Tested before and after 20 weeks intervention
  Muscle strength tested in knee extension (N)

CONTACTS AND LOCATIONS:
Overall Officials: Stig Mølsted, PhD, Principal Investigator — Department of Clinical Research, Nordsjællands Hospital, Denmark
Locations (2):
- Denmark (2):
  - Nordsjællands Hospital, Hillerød, Capital Region
  - Nordsjællands Hospital, Hillerød, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen SG, Pedersen M, Toftager-Oster JU, Saervoll CA, Fischer TK, Lindegaard B, Molsted S. Feasibility and Effects of Exercise During Working Hours in Acute Hospital Staff - A Non-Randomized Controlled Trial. J Occup Rehabil. 2025 Feb 18. doi: 10.1007/s10926-025-10275-6. Online ahead of print. PMID 39966325